CLINICAL TRIAL: NCT07282249
Title: A Multicenter, Randomized, Placebo-Controlled and Positive-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TVAX-008 Injection in the Treatment of Chronic Hepatitis B
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of TVAX-008 Injection in the Treatment of Chronic Hepatitis B
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grand Theravac Life Sciences (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YDSWX(TVAX-008)-003(III)
Record Dates: First submitted 2025-11-30; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Chronic hepatitisB

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVAX-008 and placebo (Experimental)
  Interventions: Drug: TVAV-008; Drug: Placeb
- PEG IFNα-2b (Active Comparator): PEG IFNα-2b
  Interventions: Drug: PegIFNα2b

INTERVENTIONS:
Drug: TVAV-008 — TVAV-008 will be administered per 4 weeks
  Arms: TVAX-008 and placebo
Drug: PegIFNα2b — PegIFNα will be administered per week
  Arms: PEG IFNα-2b
Drug: Placeb — Placebo will be administered per 4 weeks
  Arms: TVAX-008 and placebo

SUMMARY:
This is a multicenter, randomized, placebo-controlled (double-blind design) versus active-controlled (open-label design) Phase I clinical trial evaluating the efficacy and safety of TVAX-008 injection in subjects with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years (inclusive);
* Clinically diagnosed chronic hepatitis B (serum HBsAg positive ≥6 months);
* Subjects with a history of nucleoside (acid) analog anti-hepatitis B therapy lasting ≥6 months until screening, currently receiving antiviral therapy with a single nucleoside (acid) analog [eg, tenofovir fumarate (TAF), amitenofovir (TMF), tenofovir disoform fumarate (TDF) or entecavir (ETV), etc.], and HBV DNA<100 IU/mL within 28 days prior to the first dose of investigational product;
* Hepatitis B virus e antigen (HBeAg) negative within 28 days prior to first use of investigational product;
* HBsAg>0.05 IU/mL and HBsAg<100 IU/mL within 28 days prior to first use of investigational product;
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2× upper limit of normal (ULN) within 28 days prior to the first dose of investigational product;
* Antinuclear antibodies (ANA) negative, or abnormal but not supportive of diagnosis of autoimmune liver disease in the investigator's judgment;

Exclusion Criteria:

* Liver disease caused by other causes, including alcoholic liver disease, nonalcoholic steatohepatitis, drug-induced hepatitis, hemochromatosis, etc.;
* In addition to chronic hepatitis B, clinically important chronic diseases that, in the opinion of the investigator, make the patient unsuitable for participation in the study, including but not limited to thyroid disease requiring clinical intervention or clinically significant thyroid dysfunction, fundus disease (e.g. retinopathy), chronic lung disease with lung dysfunction, history of severe seizures or current use of antiepileptic drugs, immunodeficiency or autoimmune disease;
* Laboratory indicators or symptoms meet one or more of the following:

  1. Blood phosphorus <0.65 mmol/L;
  2. Serum albumin <35 g/L;
  3. Total bilirubin>1.5×ULN;
  4. Hemoglobin <100 g/L;
  5. Prothrombin time international normalized ratio (INR) ≥1.5;
  6. Past or present ascites, variceal bleeding, hepatorenal syndrome, hepatic encephalopathy or liver failure;Child-Pugh score B/C (see Appendix 1 for Child-Pugh classification criteria);
  7. Platelet count <125×109/L;
  8. WBC count <3×109/L;
  9. Absolute neutrophil count <1.5×109/L;
  10. Estimated glomerular filtration rate (eGFR)<50 mL/min/1.73m2[calculated using the Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI formula), see Appendix 2 for CKD-EPI formula];
  11. Imaging results show hepatocellular carcinoma, cirrhosis or liver mass (except liver cyst or hemangioma), or alpha-fetoprotein (AFP) ≥20 μg/L, or FibroScan®/FibroTouch® liver stiffness value (LSM)>10.6 kPa;
  12. Serum ceruloplasmin (CP) results suggest an increased risk of metabolic disease;
* Use of immunosuppressants within 6 months prior to first use of investigational product;
* Treatment with corticosteroids (other than topical or inhaled corticosteroids) lasting for 1 week or more within 6 months prior to first use of investigational product;
* Hepatitis C virus (HCV) antibody positive and HCV RNA positive; or hepatitis D virus (HDV) antibody positive; or human immunodeficiency virus (HIV) antibody positive; or Treponema pallidum (TP) antibody positive [except for rapid plasma reagin circular card test (RPR) or toluidine red unheated serum test (TRUST) negative];
* History of malignant tumor or recurrence within 5 years prior to the first use of investigational product;
* Previous organ transplant;
* Severe cardiac disease [including myocardial infarction, unstable angina, heart failure (New York Heart Association (NYHA) Functional Class III or IV, NYHA Functional Class criteria see Appendix 3)], renal failure, or pancreatitis;
* Diabetes mellitus with unstable drug control [glycosylated hemoglobin (HbA1c) ≥7.5%] or hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg);
* History of severe drug or food allergy;
* History of alcohol or drug abuse within 6 months prior to screening (mean alcohol consumption in ethanol: >40 g/day for men and>20 g/day for women);
* A past or current diagnosis of mental illness, especially depression or depressive tendencies;
* Use of other investigational drugs or biologics within 30 days or 5 drug half-lives (whichever is longer) prior to first use of investigational product; or participation in a clinical trial of a medical device, drug or vaccine at screening;
* Subjects who have previously taken the investigational drug TVAX-008 injection within 1 year;
* In the opinion of the investigator, participation in this trial is not appropriate due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving HBsAg lower than limit of detection (LOD) (0.05 IU/mL) and HBV DNA lower than lower limit of quantitation (LLOQ). | week72

IPD SHARING:
Plan to Share IPD: No